CLINICAL TRIAL: NCT06417229
Title: A Phase 1, Two-part, Open-label Single Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of BMS-986365, Food and Proton Pump Inhibitor Effects, and Relative Bioavailability of BMS-986365 Capsule Compared to Tablet Formulation in Healthy Adult Male Participants
Brief Title: Study to Evaluate Safety, Drug Levels, Food and Relative Bioavailability of BMS-986365 in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA228-1011
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
Keywords: BMS-986365; Pharmacokinetics; Relative Bioavailability; Healthy Male Volunteers; CC-94676; Food Effect; Proton Pump Inhibitor
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1: Cohort 1 BMS-986365 Dose 1 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Cohort 2 BMS-986365 Dose 2 Formulation 1 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Cohort 2 BMS-986365 Dose 3 Formulation 2 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Cohort 3 BMS-986365 Dose 4 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Cohort 6 BMS-986365 Dose 5 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Cohort 7 BMS-986365 Dose 6 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Cohort 8 BMS-986365 Dose 7 (Experimental)
  Interventions: Drug: BMS-986365
- Part 1: Cohort 9 BMS-986365 Dose 8 (Experimental)
  Interventions: Drug: BMS-986365
- Part 2: Cohort 4 BMS-986365 Dose 9 Fasted (Experimental)
  Interventions: Drug: BMS-986365
- Part 2: Cohort 4 BMS-986365 Dose 10 Fed (Experimental)
  Interventions: Drug: BMS-986365
- Part 2: Cohort 5 BMS-986365 Dose 11 Fasted Followed by Rabeprazole + Rabeprazole and BMS-986365 (Experimental)
  Interventions: Drug: BMS-986365; Drug: Rabeprazole

INTERVENTIONS:
Drug: BMS-986365 — Specified dose on specified days
  Other Names: CC-94676
Drug: Rabeprazole — Specified dose on specified days
  Arms: Part 2: Cohort 5 BMS-986365 Dose 11 Fasted Followed by Rabeprazole + Rabeprazole and BMS-986365

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels, food effects and relative bioavailability of BMS-986365 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male participants as determined by no clinically significant deviations from normal in medical history, physical examination, vital signs, ECGs, echocardiogram, or clinical laboratory assessments as determined by the investigator.
* Body mass index (BMI) of 18.0 to 32.0 kg/m^2, inclusive.

Exclusion Criteria:

* Any significant acute or chronic illness.
* Prior history of heart failure, ischemic heart diseases, serious cardiac arrythmias, or prolonged QT interval.
* History of allergy/hypersensitivity to any component (including excipients) of BMS-986365 study interventions or related compounds.
* Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 75
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration [AUC(0-T)] | Up to Day 75
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Up to Day 75

SECONDARY OUTCOMES:
To assess the bioavailability of BMS-986365 experimental formulation relative to the reference formulation | Up to Day 75
Incidence of adverse events (AE) | Up to Day 75
Incidence of serious adverse events (SAE) | Up to Day 75
Number of participants with physical examination abnormalities | Up to Day 75
Number of participants with vital sign abnormalities | Up to Day 75
Number of participants with clinical laboratory abnormalities | Up to Day 75
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 75

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com